CLINICAL TRIAL: NCT06883630
Title: A Phase Ib, Multi-Cohort, Open-Label, Multi-Center Clinical Trial to Evaluate the Efficacy and Safety of RC148 Injection as Monotherapy or Combination Therapy in Patients With Locally Advanced or Metastatic Non-small Cell Lung Cancer.
Brief Title: A Phase Ib Study of RC148 as Monotherapy or Combination for Locally Advanced or Metastatic NSCLC
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: RemeGen Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RC148-C002
Record Dates: First submitted 2025-03-05; First posted 2025-03-19 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin; Paclitaxel; Pemetrexed

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- AGA-, NSCLC without systemic therapy (Experimental): Combination Therapy
  Interventions: Drug: RC148 plus Carboplatin and Paclitaxel/pemetrexed
- AGA-，PD-1+, NSCLC without systemic therapy (Experimental): Monotherapy
  Interventions: Drug: RC148
- EGFR mu, Non-squamous NSCLC after EGFR-TKIs treatment (Experimental): Combination Therapy
  Interventions: Drug: RC148 plus Carboplatin and Paclitaxel/pemetrexed

INTERVENTIONS:
Drug: RC148 plus Carboplatin and Paclitaxel/pemetrexed — RC148; Carboplatin; Paclitaxel; pemetrexed
  Other Names: RC148 Injection
  Arms: AGA-, NSCLC without systemic therapy; EGFR mu, Non-squamous NSCLC after EGFR-TKIs treatment
Drug: RC148 — RC148 Monotherapy
  Other Names: RC148 Injection
  Arms: AGA-，PD-1+, NSCLC without systemic therapy

SUMMARY:
This study will evaluate the efficacy, safety, pharmacokinetics and immunogenicity of RC148 injection as a single agent or in combination for the treatment of locally advanced or metastatic non-small cell lung cancer

DETAILED DESCRIPTION:
Primary objective: to evaluate the efficacy of RC148 injection as monotherapy or combination therapy in patients locally advanced or metastatic non-small cell lung cancer;

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participate in the study and signed the ICF;
2. Be willing to and able to act on the trial and the follow up procedures;
3. Male or female, aged 18-80 years;
4. Expected survival ≥ 3 months;
5. ECOG PS score 0 or 1;
6. All participants to be enrolled in cohorts 1-5 must be diagnosed with histopathologically or cytologically confirmed, unresectable locally advanced or metastatic NSCLC (stage IIIB//IIIC/IV according to the 8th edition of UICC/AJCC) and not amendable to curative surgery or radiation as assessed by investigator.

Exclusion Criteria:

1. Histopathologically or cytologically confirmed small cell lung cancer;
2. Received major surgeries and still in recovery within 28 days before the first dose;
3. Received any live vaccine within 28 days prior to the first dose or plan to be vaccinated during the study (except for COVID-19 vaccine);
4. Received immune checkpoint inhibitor (anti-PD-1/PD-L1/CTLA-4 antibody) or other immune checkpoint inhibitor treatment within 28 days prior to the first dose, or experienced prior permanent immunotherapy discontinuation due to immunotoxicity;
5. Participated in other clinical trials and received other investigational anti-tumor therapy within 28 days prior to the first dose;
6. Poor compliance and unable to complete the study procedures as assessed by investigator;
7. Have any other medical conditions, abnormal physical examinations or laboratory examinations that would be suspected interfere with participation or evaluation of the trial or increase the risk to the participant, in view of the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-03-13 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 24 months
  Tumor assessment will be performed until radiographic disease progression, initiation of new anticancer therapy, withdrawal of consent, death, loss to follow-up, or other end of study criterion is met, whichever is earlier.

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | 24 months
  Tumor assessment will be performed until radiographic disease progression, initiation of new anticancer therapy, withdrawal of consent, death, loss to follow-up, or other end of study criterion is met, whichever is earlier.
Duration of Response (DOR) | 24 months
  Tumor assessment will be performed until radiographic disease progression, initiation of new anticancer therapy, withdrawal of consent, death, loss to follow-up, or other end of study criterion is met, whichever is earlier.
Progression-free survival (PFS) | 24 months
  Tumor assessment will be performed until radiographic disease progression, initiation of new anticancer therapy, withdrawal of consent, death, loss to follow-up, or other end of study criterion is met, whichever is earlier.
Overall survival (OS) | 24 months
  Tumor assessment will be performed until radiographic disease progression, initiation of new anticancer therapy, withdrawal of consent, death, loss to follow-up, or other end of study criterion is met, whichever is earlier.
Number of participants with adverse events (AEs) | 24 months
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment.
Incidence of RC148 anti-drug antibody (ADA) | 24 months
  Serum samples will be collected from participants for ADA analysis of RC148. The blood sampling time points and time windows are described in protocol
Maximum observed concentration (Cmax) of RC148 | 24 months
  Serum concentrations of RC148 in individual subjects at different time points after RC148 administration

CONTACTS AND LOCATIONS:
Overall Officials: li zhang, Study Director — Sun Yat-sen University
Locations (24):
- China (24):
  - Beijing Tiantan Hospital of Capital Medical University, Beijing, Beijing Municipality
  - Peking University Cancer Hospital, Beijing, Beijing Municipality
  - Shunde Hospital of Southern Medical University, Foshan, Guangdong
  - The First People's Hospital of Shunde, Foshan, Guangdong
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - The First affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Jiangmen Central Hospital, Jiangmen, Guangdong
  - The Second Affiliated Hospital of Guilin Medical College, Gulin, Guangxi
  - Affiliated Cancer Hospital of Guangxi Medical University, Nanning, Guangxi
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Nanyang Second General Hospital, Hanyang, Henan
  - The First Affiliated Hospital of Xinxiang Medical College, Xinxiang, Henan
  - Henan cancer hospital, Zhengzhou, Henan
  - Union Hospital Tongji Medical College Huazhong University Of Science And Technologe, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Binzhou Medical University Hospital, Binzhou, Shandong
  - Jinan Central Hospital, Jinan, Shandong
  - Linyi Cancer Hospital, Linyi, Shandong
  - Tianjin Medical University Cancer Institute Hospital, Tianjin, Tianjin Municipality
  - Yunnan Cancer Hospital, Kunming, Yunnan
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Taizhou Hospital of Zhejiang Province, Taizhou, Zhejiang